CLINICAL TRIAL: NCT03869658
Title: Food Talk: A New App for Daily Food Monitoring
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Susan Roberts, Senior Scientist and Lab Director, Tufts University
Other Study IDs: 1234
Record Dates: First submitted 2018-09-19; First posted 2019-03-11 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Dietary Intake
Keywords: Voice recognition; 24-hr diet recall; Mobile application; Self-report

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: COCO application — All participants will complete a screening survey to determine their eligibility for the study, if eligible and willing to participate, he or she will sign an informed consent form. Once participants are enrolled in the study, a demographics questionnaire will be completed along with 5 days of food tracking on the COCO application. Between days 3 and 7, participants will complete two 24-hr diet recall, one a day, and a patient satisfaction questionnaire.

SUMMARY:
This project will pilot test a new app for self-monitoring food intake using natural spoken language (by voice recognition or text) to provide daily estimates of energy and nutrient intakes with a phone app.

DETAILED DESCRIPTION:
Self-recording food intake is recommended for weight management and healthy eating. However, current methods, including web platforms and apps, are often burdensome leading to short-term use by the consumer. The solution uses cutting-edge speech and language understanding technology to streamline the food logging process. With this technology, the user simply describes what they ate and the system automatically selects the appropriate items and quantities consumed from the USDA food database, which calculates the nutrition profile of the entry.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy men and women 18-65 years if age
* Currently participating in ongoing studies at the HNRCA
* Willing and able to sign written informed consent prior to study entry
* iPhone (iOS 11 or higher) user willing to download the COCO application and record food intake for 5 days

Exclusion Criteria:

* Android or iPhone (iOs 10 or lower) user unable to download and use the COCO application
* Holds a graduate degree in nutrition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be recruited from the local community around Boston, Massachusetts. Recruitment methods include posting flyers, social and local media advertisements, word of mouth, and emails to HNRCA mailing lists.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in energy intake using food application COCO | Between days 3 and 7 of the study
  The primary outcome will be to assess whether food capture using the mobile application is comparable with conventional 24-hour dietary recall. This will be done by measuring the energy intake (mean of two days) in the two methods.
Change in energy intake using 24 hour dietary recall | Between days 3 and 7 of the study
  The primary outcome will be to assess whether food capture using the mobile application is comparable with conventional 24-hour dietary recall. This will be done by measuring the energy intake (mean of two days) in the two methods.

SECONDARY OUTCOMES:
Accuracy of food capture method using mobile application | Between days 3 and 7 of the study
  The secondary outcome will measure the energy and nutrient content reported by the mobile application over time. Measured energy intake in a subset of participants in another study that provides dietary intake data will be compared to food intake data using the mobile application.

OTHER OUTCOMES:
Application feasibility | Betweens days 5 and 7
  Feasibility of the use of the application to record dietary intake will be measured through a patient satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Beydoun MA. The obesity epidemic in the United States--gender, age, socioeconomic, racial/ethnic, and geographic characteristics: a systematic review and meta-regression analysis. Epidemiol Rev. 2007;29:6-28. doi: 10.1093/epirev/mxm007. Epub 2007 May 17. PMID 17510091
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Finkelstein EA, Trogdon JG, Cohen JW, Dietz W. Annual medical spending attributable to obesity: payer-and service-specific estimates. Health Aff (Millwood). 2009 Sep-Oct;28(5):w822-31. doi: 10.1377/hlthaff.28.5.w822. Epub 2009 Jul 27. PMID 19635784